CLINICAL TRIAL: NCT01220856
Title: A Phase 2 Multicenter, Randomized, Open Label, Parallel Assignment, Pilot Study to Assess the Efficacy and Safety of Reparixin Following Islet Transplantation in Patients With Type 1 Diabetes Mellitus
Brief Title: Reparixin in Pancreatic Islet Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REP0110; 2010-019424-31 (EudraCT Number)
Record Dates: First submitted 2010-10-07; First posted 2010-10-14 (Estimated); Results first posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-02

CONDITIONS: Pancreatic Islet Transplantation in Type 1 Diabetes Mellitus
Keywords: Islet transplantation; Type 1 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — reparixin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reparixin (Experimental): Reparixin + Immunosuppression
  Reparixin was administered at a dose of 2.772 mg/kg body weight/hour for 7 days (168 hours) at each transplant. It was administered as a continuous IV infusion into a (high-flow) central vein. Investigational Product infusion was to begin approximately 12 hours (range between 6 to 16 hours) before each pancreatic islet infusion was started. The Investigator identified the time to start study drug administration.
  Reparixin was given to all patients of this arm using the same dosing solution (reparixin 11.00 mg/mL), but the pump rate was adjusted to provide an infusion rate of approximately 0.25 mL/kg/hour.
  For immunosoppression regimen see the other arm description.
  Interventions: Drug: Reparixin
- No experimental intervention (No Intervention): Immunosuppression only. Induction: First islet infusion: anti-thymocyte globulin (ATG), administered IV (central vein) at the dose of 1.5 mg/kg on Day -1, 0, 1, and 2 of islet infusion. The first ATG injection was preceded by a bolus IV injection of 500 mg methylprednisolone. Induction for the second islet infusion was to be administered per center practice. Maintenance: Mycophenolate mofetil (MMF), administered orally at the dose of 1 g twice a day, starting on Day -1 of the first islet infusion; Tacrolimus, administered orally starting on Day -1 of the first islet infusion at a dose of 0.087 mg/kg twice a day. Thereafter, dosing was to be targeted to blood trough levels of 8 to 10 ng/mL. Administration continued up to Month 3 after the first transplant. Rapamycin was to replace tacrolimus from Month 3 after the first transplant. It was to be administered orally at the starting dose of 0.1 mg/kg once a day, then targeted to a blood trough level of 10 to 12 ng/mL.

INTERVENTIONS:
Drug: Reparixin — Reparixin + immunosuppression
  Other Names: REP
  Arms: Reparixin

SUMMARY:
Inhibition of CXCL8 activity might represent a relevant therapeutic target to prevent injury occurring after pancreatic islet transplantation. Reparixin is a novel and specific inhibitor of CXCL8. This study is designed to explore the efficacy of reparixin in preventing graft dysfunction after islet transplantation in type 1 diabetes patients (T1D).

DETAILED DESCRIPTION:
Pancreatic islet transplantation has become a feasible option in the treatment of T1D which offers advantages over whole pancreas transplantation. However to date insulin independence can be obtained in most cases only after the patient has received repeated infusions from several donors. A non-specific immune response, mediated predominantly by innate inflammatory processes, coupled with specific cellular immune responses, possibly promoted by early inflammation, play a major role in the loss of transplanted islets from the liver. PMNs have been found to be the predominant cell types infiltrating in vitro the islets. In this regard, CXCL8 has been shown to be expressed by human islets and could play a crucial role in triggering the inflammatory reaction. Thus, CXCL8 might represent a relevant therapeutic target to prevent early graft failure. The efficacy of reparixin in improving graft outcome in mice models of intrahepatic islet transplantation, as well as the safety shown in human phase 1 and 2 studies, provide a rationale for a clinical study aimed at evaluating the effect of reparixin in preventing graft dysfunction after islet transplantation in T1D patients.

ELIGIBILITY:
Inclusion criteria:

* Ages 18-65 years, inclusive.
* Patients eligible for pancreatic islet transplantation based on local accepted practice and guidelines. This includes at least: a)clinical history compatible with T1D with insulin-dependence for >5 years; b) undetectable stimulated (arginine or MMTT) C-peptide levels (<0.3 ng/mL) in the 12 months before transplant. Sites will comply with any additional or more stringent criteria locally accepted, as per centre practice.
* Patients with adequate renal reserve as per calculated creatinine clearance (CLcr) > 60 mL/min according to the Cockcroft-Gault formula (1976).
* Planned intrahepatic islet transplantation alone from a non-living donor with brain death.
* Planned infusion of 4000 to 7000 islet equivalent (IEQ)/kg body weight.
* Patients willing and able to comply with the protocol procedures for the duration of the study, including scheduled follow-up visits and examinations.
* Patients given written informed consent, prior to any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.

Exclusion criteria:

* Recipients of any previous transplant, except from recipients of a previous pancreatic islet transplantation that has failed, are off immunosuppression since at least 1 year and have negative anti-HLA.
* Recipients of islet from a non-heart beating donor.
* A body mass index >30 kg/m2 or patient weight <45 kg.
* Pre-transplant average daily insulin requirement >1 IU/kg/day.
* Pre-transplant HbA1c >11%.
* Patients with hepatic dysfunction as defined by increased ALT/AST > 3 x ULN and increased total bilirubin > 3mg/dL [>51.3 micromol/L]).
* Patients who receive treatment for a medical condition requiring chronic use of systemic steroids.
* Treatment with any anti-diabetic medication other than insulin within 4 weeks of transplant.
* Use of any investigational agent within 4 weeks of enrolment.
* Hypersensitivity to:

  * ibuprofen or to more than one non steroidal anti-inflammatory drug
  * medications belonging to the class of sulfonamides, such as sulfamethazine, sulfamethoxazole, sulfasalazine, nimesulide or celecoxib.
* Pregnant or breast-feeding women; unwillingness to use effective contraceptive measures (females and males).

Sites will comply with any additional exclusion criteria locally accepted, as per centre practice.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-07-28 (Actual); Primary Completion 2013-04-30 (Actual); Study Completion 2013-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Piemonti, MD, Principal Investigator — Fondazione Centro San Raffaele del Monte Tabor - Milan; Italy; Barbara Ludwig, MD, Principal Investigator — University Hospital Carl Gustav Carus - Dresden; Germany
Locations (2):
- University Hospital Carl Gustav Carus Dresden, Dresden, Germany
- Ospedale San Raffaele, Milan, Italy

REFERENCES:
- [Derived] Ajmal N, Bogart MC, Khan P, Max-Harry IM, Healy AM, Nunemaker CS. Identifying Promising Immunomodulators for Type 1 Diabetes (T1D) and Islet Transplantation. J Diabetes Res. 2024 Dec 20;2024:5151171. doi: 10.1155/jdr/5151171. eCollection 2024. PMID 39735417
- [Derived] Citro A, Cantarelli E, Piemonti L. Anti-inflammatory strategies to enhance islet engraftment and survival. Curr Diab Rep. 2013 Oct;13(5):733-44. doi: 10.1007/s11892-013-0401-0. PMID 23912763

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 9 patients were enrolled into the study; 6 were randomized to reparixin and 3 to the control group. All in the control group and 2 in the reparixin group were withdrawn after Transplant 1 due to graft loss. 4 in the reparixin group received Transplant 2. Thereafter, 1 was withdrawn due to graft loss. 1 was lost to follow-up.
Groups:
- Reparixin: Reparixin + Immunosuppression
  Reparixin was administered at a dose of 2.772 mg/kg body weight/hour for 7 days (168 hours) at each transplant. It was administered as a continuous IV infusion into a (high-flow) central vein. Investigational Product infusion was to begin approximately 12 hours (range between 6 to 16 hours) before each pancreatic islet infusion was started. The Investigator identified the time to start study drug administration.
  Reparixin was given to all patients of this arm using the same dosing solution (reparixin 11.00 mg/mL), but the pump rate was adjusted to provide an infusion rate of approximately 0.25 mL/kg/hour.
  For immunosuppression regimen see the other arm description.
  Reparixin: Reparixin + immunosuppression
Period: Overall Study
Arm/Group | Reparixin | No Experimental Intervention
Started | 6 | 3
Completed | 2 | 0
Not Completed | 4 | 3
Not completed — graft loss | 3 | 3
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: All patients who were randomized into the study were included in the safety population.
Groups:
- Reparixin: Reparixin + Immunosuppression
  Reparixin was administered at a dose of 2.772 mg/kg body weight/hour for 7 days (168 hours) at each transplant. It was administered as a continuous IV infusion into a (high-flow) central vein. Investigational Product infusion was to begin approximately 12 hours (range between 6 to 16 hours) before each pancreatic islet infusion was started. The Investigator identified the time to start study drug administration.
  Reparixin was given to all patients of this arm using the same dosing solution (reparixin 11.00 mg/mL), but the pump rate was adjusted to provide an infusion rate of approximately 0.25 mL/kg/hour.
  For immunosoppression regimen see the other arm description.
  Reparixin: Reparixin + immunosuppression
- Total: Total of all reporting groups
Arm/Group | Reparixin | No Experimental Intervention | Total
Number analyzed (Participants) | 6 | 3 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 9
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (8.8) | 48.0 (7.0) | 46.8 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  Italy | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Insulin-independent Patients Following Single Infusion Islet Cell Transplantation at Day 75 +/- 5
Description: Insulin-independence was defined as freedom from the need to take exogenous insulin for 14 or more consecutive days, with adequate glycemic control, as defined by:
  * HbA1c level of less than 7%;
  * glucose level after an overnight fast not exceeding 140 mg/dL (7.8 mmol/L) more than 3 times a week (based on measuring capillary glucose level a minimum of 7 times in a 7-day period);
  * glucose level not exceeding 2-hour postprandial levels of 180 mg/dL (10 mmol/L) more than 4 times a week (based on measuring capillary glucose level a minimum of 21 times in a 7-day period).
Time Frame: day 75 +/- 5 post-transplant
Population: Efficacy Population: All patients who were randomized and received the transplant were included in the efficacy population.
Measure: Number; unit: percentage of patients
Arm/Group | Reparixin | No Experimental Intervention
Number analyzed (Participants) | 6 | 3
percentage of patients | 0 | 0

2. Other Pre Specified Outcome: The Percentage of Insulin-independent Patients Following Islet Cell Transplantation up to One Year After the Last Transplant
Description: as for outcome 1
Time Frame: up to one year after the transplant
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Reparixin | No Experimental Intervention
Number analyzed (Participants) | 6 | 3
percentage of patients
  transplant 1 | 0 | 0
  transplant 2: number analyzed (Participants) | 4 | 0
  transplant 2 | 50 |

3. Other Pre Specified Outcome: Time to Achieve Insulin-independence After the Transplant 2
Description: Time to achieve insulin-independence after the transplant was defined as the number of days between islet infusion and onset of insulin-independence. This was calculated as: date of onset of insulin-independence minus the islet infusion date.
Time Frame: up to 1 year after transplant 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Reparixin | No Experimental Intervention
Number analyzed (Participants) | 3 | 0
days | 66.3 (73.7) |

4. Other Pre Specified Outcome: Total Time of Insulin Independence After the Transplant
Description: Total time of insulin-independence after the transplant. This was defined as the number of days between the onset and loss of insulin-independence and was calculated as the date of loss of insulin-independence minus the date of onset of insulin-independence.
  Of the 3 patients who achieve insulin-independence after transplant 2, only 2 remained insulin-independent up to 1 year and the mean (SD) total time of insulin-independence after the second transplant was 276 (96.2) days with a range between 208 and 344 days.
Time Frame: up to 1 year after transplant 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: total number of days
Arm/Group | Reparixin | No Experimental Intervention
Number analyzed (Participants) | 2 | 0
total number of days | 276.0 (96.2) |

5. Other Pre Specified Outcome: Absolute Change in Average Daily Insulin Requirements From Pre-transplant Levels
Description: Daily insulin requirement was calculated as the average requirement over the previous week (seven days).
Time Frame: Months 1, 3, 6, 12 post-transplant
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/kg/day
Arm/Group | Reparixin | No Experimental Intervention
Number analyzed (Participants) | 6 | 3
IU/kg/day
  Month 1 (transplant 1) | -0.3 (0.3) | 0.1 (0.1)
  Month 3 (transplant 1): number analyzed (Participants) | 4 | 0
  Month 3 (transplant 1) | -0.3 (0.2) |
  Month 6 (transplant 1): number analyzed (Participants) | 3 | 0
  Month 6 (transplant 1) | -0.2 (0.0) |
  Month 1 (transplant 2): number analyzed (Participants) | 4 | 0
  Month 1 (transplant 2) | -0.6 (0.2) |
  Month 3 (transplant 2): number analyzed (Participants) | 4 | 0
  Month 3 (transplant 2) | -0.6 (0.3) |
  Month 6 (transplant 2): number analyzed (Participants) | 4 | 0
  Month 6 (transplant 2) | -0.5 (0.4) |
  Month 12 (transplant 2): number analyzed (Participants) | 2 | 0
  Month 12 (transplant 2) | -0.7 (0.4) |

6. Other Pre Specified Outcome: Percentage Change in Average Daily Insulin Requirements From Pre-transplant Levels
Description: Daily insulin requirement was calculated as the average requirement over the previous week (seven days).
Time Frame: Months 1, 3, 6, 12 post-transplant
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Reparixin | No Experimental Intervention
Number analyzed (Participants) | 6 | 3
Percentage change
  Month 1 (transplant 1) | -41.9 (39.9) | 16.4 (20.2)
  Month 3 (transplant 1): number analyzed (Participants) | 4 | 0
  Month 3 (transplant 1) | -50.3 (24.4) |
  Month 6 (transplant 1): number analyzed (Participants) | 3 | 0
  Month 6 (transplant 1) | -32.0 (8.9) |
  Month 1 (transplant 2): number analyzed (Participants) | 4 | 0
  Month 1 (transplant 2) | -90.8 (11.3) |
  Month 3 (transplant 2): number analyzed (Participants) | 4 | 0
  Month 3 (transplant 2) | -88.7 (17.8) |
  Month 6 (transplant 2): number analyzed (Participants) | 4 | 0
  Month 6 (transplant 2) | -81.8 (36.5) |
  Month 12 (transplant 2): number analyzed (Participants) | 2 | 0
  Month 12 (transplant 2) | -100.0 (0.0) |

7. Other Pre Specified Outcome: Absolute Change in Fasted HbA1c From Pre-transplant Levels
Description: The absolute change between the time-point value and baseline value.
Time Frame: Months 1, 3, 6, 12 post-transplant
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of Hb
Arm/Group | Reparixin | No Experimental Intervention
Number analyzed (Participants) | 6 | 3
Percentage of Hb
  Month 1 (transplant 1) | -1.53 (0.49) | -0.87 (0.40)
  Month 3 (transplant 1): number analyzed (Participants) | 4 | 0
  Month 3 (transplant 1) | -2.90 (0.74) |
  Month 6 (transplant 1): number analyzed (Participants) | 3 | 0
  Month 6 (transplant 1) | -1.87 (0.60) |
  Month 1 (transplant 2): number analyzed (Participants) | 4 | 0
  Month 1 (transplant 2) | -3.15 (0.57) |
  Month 3 (transplant 2): number analyzed (Participants) | 4 | 0
  Month 3 (transplant 2) | -3.10 (0.76) |
  Month 6 (transplant 2): number analyzed (Participants) | 4 | 0
  Month 6 (transplant 2) | -3.05 (1.03) |
  Month 12 (transplant 2): number analyzed (Participants) | 2 | 0
  Month 12 (transplant 2) | -3.65 (0.92) |

8. Other Pre Specified Outcome: Percentage Change in Fasted HbA1c From Pre-transplant Levels
Description: The absolute percentage between the time-point value and baseline value.
Time Frame: Months 1, 3, 6, 12 post-transplant
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Reparixin | No Experimental Intervention
Number analyzed (Participants) | 6 | 3
Percentage change
  Month 1 (transplant 1) | -16.7 (4.5) | -11.2 (5.4)
  Month 3 (transplant 1): number analyzed (Participants) | 4 | 0
  Month 3 (transplant 1) | -30.3 (7.9) |
  Month 6 (transplant 1): number analyzed (Participants) | 3 | 0
  Month 6 (transplant 1) | -19.7 (7.2) |
  Month 1 (transplant 2): number analyzed (Participants) | 4 | 0
  Month 1 (transplant 2) | -32.8 (5.9) |
  Month 3 (transplant 2): number analyzed (Participants) | 4 | 0
  Month 3 (transplant 2) | -32.2 (7.4) |
  Month 6 (transplant 2): number analyzed (Participants) | 4 | 0
  Month 6 (transplant 2) | -31.6 (10.1) |
  Month 12 (transplant 2): number analyzed (Participants) | 2 | 0
  Month 12 (transplant 2) | -37.4 (9.2) |

9. Other Pre Specified Outcome: The Percentage of Patients Free of Hypoglycaemic Events With Reduced Awareness
Description: Reduced awareness is defined as a reduced ability to recognize symptoms of hypoglycemia, sometimes referred to as "hypoglycemia unawareness".
Time Frame: Months 1, 3, 6, 12 post-transplant
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Reparixin | No Experimental Intervention
Number analyzed (Participants) | 6 | 3
Percentage of patients
  month 1 (transplant 1) | 100 | 100
  month 3 (transplant 1): number analyzed (Participants) | 4 | 0
  month 3 (transplant 1) | 100 |
  month 6 (transplant 1): number analyzed (Participants) | 3 | 0
  month 6 (transplant 1) | 100 |
  month 1 (transplant 2): number analyzed (Participants) | 4 | 0
  month 1 (transplant 2) | 100 |
  month 3 (transplant 2): number analyzed (Participants) | 4 | 0
  month 3 (transplant 2) | 100 |
  month 6 (transplant 2): number analyzed (Participants) | 4 | 0
  month 6 (transplant 2) | 100 |
  month 12 (transplant 2): number analyzed (Participants) | 2 | 0
  month 12 (transplant 2) | 100 |

10. Other Pre Specified Outcome: Number of Participants With Adverse Events by Severity and With Serious Adverse Events
Description: Safety was assessed by monitoring the incidence and severity of adverse events (AEs) and serious AEs (SAEs) throughout the study up to 1 year after last transplant.
  A serious adverse event is an adverse reaction that results in death, is life-threatening, requires hospitalisation or prolongation of existing hospitalisation, results in persistent or significant disability or incapacity, or is a birth defect.
Time Frame: up to 1 year after transplant
Population: Safety Population: all patients who were randomized into the study.
Measure: Number; unit: participants
Arm/Group | Reparixin | No Experimental Intervention
Number analyzed (Participants) | 6 | 3
participants
  TEAE mild | 5 | 2
  TEAE moderate | 6 | 2
  TEAE severe | 3 | 1
  SAE | 3 | 1

11. Other Pre Specified Outcome: AUC (-10 to 120 Minutes Post-dose) of Glucose Derived From Mixed Meal Tolerance Test (MMTT) at 1, 3, 6 and 12 Months Post-transplant
Description: Glucose level reflects the metabolic control. The MMTT was performed after an overnight fast, at baseline (within 1 week prior to randomization), and at each of the following timepoints.
  AUC was calculated using the trapezoidal rule.
Time Frame: -10 to 120 Minutes Post-dose at Months 1, 3, 6, 12 post-transplant
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg*hr/dL
Arm/Group | Reparixin | No Experimental Intervention
Number analyzed (Participants) | 6 | 3
mg*hr/dL
  Month 1, transplant 1 | 318.9 (155.1) | 308.3 (105.4)
  Month 3, transplant 1: number analyzed (Participants) | 4 | 0
  Month 3, transplant 1 | 235.0 (77.6) |
  Month 6, transplant 1: number analyzed (Participants) | 3 | 0
  Month 6, transplant 1 | 277.2 (59.9) |
  Month 1, transplant 2: number analyzed (Participants) | 4 | 0
  Month 1, transplant 2 | 162.5 (36.3) |
  Month 3, transplant 2: number analyzed (Participants) | 4 | 0
  Month 3, transplant 2 | 171.2 (58.1) |
  Month 6, transplant 2: number analyzed (Participants) | 4 | 0
  Month 6, transplant 2 | 184.1 (74.4) |
  Month 12, last transplant: number analyzed (Participants) | 2 | 0
  Month 12, last transplant | 123.7 (18.3) |

12. Other Pre Specified Outcome: AUC (-10 to 120 Minutes Post-dose) of C-peptide Derived From Mixed Meal Tolerance Test (MMTT) at 1, 3, 6 and 12 Months Post-transplant
Description: C-peptide level is an indirect measure of pancreatic beta-cell function. The MMTT was performed after an overnight fast, at baseline (within 1 week prior to randomization), and at each of the following timepoints.
  AUC was calculated using the trapezoidal rule.
Time Frame: -10 to 120 Minutes Post-dose at Months 1, 3, 6, 12 post-transplant
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg*hr/dL
Arm/Group | Reparixin | No Experimental Intervention
Number analyzed (Participants) | 6 | 3
mg*hr/dL
  Month 1 (transplant 1) | 0.951 (0.875) | 0.200 (0.000)
  Month 3 (transplant 1): number analyzed (Participants) | 4 | 0
  Month 3 (transplant 1) | 1.789 (1.059) |
  Month 6 (transplant 1): number analyzed (Participants) | 3 | 0
  Month 6 (transplant 1) | 1.426 (1.114) |
  Month 1 (transplant 2): number analyzed (Participants) | 4 | 0
  Month 1 (transplant 2) | 3.302 (1.661) |
  Month 3 (transplant 2): number analyzed (Participants) | 4 | 0
  Month 3 (transplant 2) | 2.488 (2.038) |
  Month 6 (transplant 2): number analyzed (Participants) | 4 | 0
  Month 6 (transplant 2) | 2.531 (1.831) |
  Month 12 (last transplant): number analyzed (Participants) | 2 | 0
  Month 12 (last transplant) | 4.042 (1.683) |

13. Other Pre Specified Outcome: AUC (-10 to 120 Minutes Post-dose) of Insulin Derived From Mixed Meal Tolerance Test (MMTT) at 1, 3, 6 and 12 Months Post-transplant
Description: Insulin level is a direct measure of pancreatic beta-cell function. The MMTT was performed after an overnight fast, at baseline (within 1 week prior to randomization), and at each of the following timepoints.
  AUC was calculated using the trapezoidal rule.
Time Frame: -10 to 120 Minutes Post-dose at Months 1, 3, 6, 12 post-transplant
Population: Efficacy Population: All patients who were randomized and received the transplant were included in the efficacy population. This population was based on the treatment randomized, regardless of the treatment actually received.
Measure: Mean (Standard Deviation); unit: μU*hr/mL
Arm/Group | Reparixin | No Experimental Intervention
Number analyzed (Participants) | 6 | 3
μU*hr/mL
  Month 1 (transplant 1) | 19.08 (15.72) | 7.58 (2.91)
  Month 3 (transplant 1): number analyzed (Participants) | 4 | 0
  Month 3 (transplant 1) | 28.25 (33.43) |
  Month 6 (transplant 1): number analyzed (Participants) | 3 | 0
  Month 6 (transplant 1) | 13.41 (7.81) |
  Month 1 (transplant 2): number analyzed (Participants) | 4 | 0
  Month 1 (transplant 2) | 20.99 (11.89) |
  Month 3 (transplant 2): number analyzed (Participants) | 4 | 0
  Month 3 (transplant 2) | 22.85 (23.07) |
  Month 6 (transplant 2): number analyzed (Participants) | 4 | 0
  Month 6 (transplant 2) | 19.97 (16.40) |
  Month 12 (transplant 2): number analyzed (Participants) | 2 | 0
  Month 12 (transplant 2) | 36.04 (13.83) |

14. Other Pre Specified Outcome: AUC(-10 to 120 Min Post Dose)/IEQ/kg for C Peptide Derived From Mixed Meal Tolerance Test (MMTT) at 1, 3, 6 Months Post-transplant 1
Description: For Transplant 1 (patients on reparixin), the mean C-Peptide AUC (derived from the MMTT) corrected by IEQ/kg values were calculated.
  AUC was calculated using the trapezoidal rule and normalized by the actual number of islet equivalents (IEQ) per kilo infused (IEQ/kg).
Time Frame: -10 to 120 Minutes Post-dose at Months 1, 3, 6, 12 post-transplant
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: (mg*hr/dL)/IEQ/kg
Arm/Group | Reparixin | No Experimental Intervention
Number analyzed (Participants) | 6 | 3
(mg*hr/dL)/IEQ/kg
  Month 1 (transplant 1) | 0.193 (0.158) | 0.044 (0.004)
  Month 3 (transplant 1): number analyzed (Participants) | 4 | 0
  Month 3 (transplant 1) | 0.366 (0.158) |
  Month 6 (transplant 1): number analyzed (Participants) | 3 | 0
  Month 6 (transplant 1) | 0.341 (0.265) |

15. Other Pre Specified Outcome: The Percentage of Patients Free of Severe Hypoglycaemic Events
Description: A severe hypoglycemic event is defined as an event with one of the following symptoms: "memory loss, confusion, uncontrollable behavior, irrational behavior, unusual difficulty in awakening, suspected seizure, seizure, loss of consciousness, or visual symptoms", in which the subject was unable to treat him/herself and which was associated with either a blood glucose level <54mg/dL or prompt recovery after oral carbohydrate, i.v. glucose, or glucagon administration.
Time Frame: Months 1, 3, 6, 12 post-transplant
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Reparixin | No Experimental Intervention
Number analyzed (Participants) | 6 | 3
Percentage of patients
  month 1 (transplant 1) | 100 | 100
  month 3 (transplant 1): number analyzed (Participants) | 4 | 0
  month 3 (transplant 1) | 100 |
  month 6 (transplant 1): number analyzed (Participants) | 3 | 0
  month 6 (transplant 1) | 100 |
  month 1 (transplant 2): number analyzed (Participants) | 4 | 0
  month 1 (transplant 2) | 100 |
  month 3 (transplant 2): number analyzed (Participants) | 4 | 0
  month 3 (transplant 2) | 100 |
  month 6 (transplant 2): number analyzed (Participants) | 4 | 0
  month 6 (transplant 2) | 100 |
  month 12 (transplant 2): number analyzed (Participants) | 2 | 0
  month 12 (transplant 2) | 100 |

16. Other Pre Specified Outcome: Beta-cell Function as Assessed by Beta-score
Description: The beta-score provides a simple clinical scoring system that encompasses glycemic control, diabetes therapy, and endogenous insulin secretion that correlates well with physiological measures of beta-cell function. On this basis, it is suitable as an overall measure of beta-cell transplant function.
  Beta score is a composite scoring system based on fasting plasma glucose values, HbA1c, insulin independence or use of insulin/OHAs, and the determination of stimulated C-peptide levels. Normal values are given a score of 2, intermediate values merit a score of 1, and clearly abnormal values garner no points. Thus, a perfect score is 8, and a score of 0 indicates absolute absence of beta-cell function.
Time Frame: Months 1, 3, 6, 12 post-transplant
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reparixin | No Experimental Intervention
Number analyzed (Participants) | 6 | 3
score on a scale
  Month 1, transplant 1 | 1.83 (1.17) | 1.33 (1.53)
  Month 3, transplant 1: number analyzed (Participants) | 4 | 0
  Month 3, transplant 1 | 3.75 (1.26) |
  Month 6, transplant 1: number analyzed (Participants) | 3 | 0
  Month 6, transplant 1 | 1.67 (1.53) |
  Month 1, transplant 2: number analyzed (Participants) | 4 | 0
  Month 1, transplant 2 | 5.25 (1.50) |
  Month 3, transplant 2: number analyzed (Participants) | 4 | 0
  Month 3, transplant 2 | 4.75 (1.89) |
  Month 6, transplant 2: number analyzed (Participants) | 4 | 0
  Month 6, transplant 2 | 4.75 (2.63) |
  Month 12, transplant 2: number analyzed (Participants) | 2 | 0
  Month 12, transplant 2 | 6.50 (0.71) |

17. Other Pre Specified Outcome: Beta-cell Function as Assessed by TEF/IEQ/kg Ratio
Description: The TEF/IEQ/kg ratio is a parameter to assess transplant efficiency corrected by the number of transplanted islets.
Time Frame: At months 1, 3, 6 after transplant 1 and months 1,3, 6, and 12 after transplant 2
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Reparixin | No Experimental Intervention
Number analyzed (Participants) | 6 | 3
ratio
  Month 1 (transplant 1) | 111.9 (64.1) | 13.6 (49.6)
  Month 3 (transplant 1): number analyzed (Participants) | 4 | 0
  Month 3 (transplant 1) | 176.6 (105.0) |
  Month 6 (transplant 1): number analyzed (Participants) | 3 | 0
  Month 6 (transplant 1) | 121.1 (30.0) |
  Month 1 (transplant 2): number analyzed (Participants) | 4 | 0
  Month 1 (transplant 2) | 1.143 (0.278) |
  Month 3 (transplant 2): number analyzed (Participants) | 4 | 0
  Month 3 (transplant 2) | 1.133 (0.336) |
  Month 6 (transplant 2): number analyzed (Participants) | 4 | 0
  Month 6 (transplant 2) | 1.100 (0.407) |
  Month 12 (transplant 2): number analyzed (Participants) | 2 | 0
  Month 12 (transplant 2) | 1.320 (0.212) |

18. Other Pre Specified Outcome: Serum Level of Alanine Amino Transferase (ALT)
Description: ALT is commonly measured clinically as part of liver function tests.
Time Frame: Pre-transplant and at days 1-7 and months 1 and 3 post-transplant
Population: Safety population: all patients who were randomized into the study.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Reparixin | No Experimental Intervention
Number analyzed (Participants) | 6 | 3
U/L
  Pre-transplant 1 | 23.0 (9.0) | 28.7 (22.9)
  Day 1 post-transplant 1 | 27.5 (8.7) | 24.7 (18.6)
  Day 2 post-transplant 1 | 26.3 (9.3) | 36.3 (29.7)
  Day 3 post-transplant 1 | 29.7 (9.7) | 46.3 (34.9)
  Day 4 post-transplant 1 | 38.5 (9.0) | 64.7 (23.0)
  Day 5 post-transplant 1 | 63.7 (21.9) | 98.0 (33.2)
  Day 6 post-transplant 1 | 86.0 (34.0) | 108.3 (34.4)
  Day 7 post-transplant 1: number analyzed (Participants) | 5 | 3
  Day 7 post-transplant 1 | 114.6 (56.4) | 108.3 (45.7)
  Month 1 (transplant 1) | 25.8 (7.7) | 29.7 (28.9)
  Month 3 (transplant 1): number analyzed (Participants) | 4 | 0
  Month 3 (transplant 1) | 25.0 (8.7) |
  Pre-transplant 2: number analyzed (Participants) | 4 | 0
  Pre-transplant 2 | 18.5 (7.9) |
  Day 1 post-transplant 2: number analyzed (Participants) | 4 | 0
  Day 1 post-transplant 2 | 24.8 (10.8) |
  Day 2 post-transplant 2: number analyzed (Participants) | 4 | 0
  Day 2 post-transplant 2 | 22.8 (9.3) |
  Day 3 post-transplant 2: number analyzed (Participants) | 4 | 0
  Day 3 post-transplant 2 | 22.8 (7.5) |
  Day 4 post-transplant 2: number analyzed (Participants) | 4 | 0
  Day 4 post-transplant 2 | 28.8 (10.8) |
  Day 5 post-transplant 2: number analyzed (Participants) | 4 | 0
  Day 5 post-transplant 2 | 31.8 (11.7) |
  Day 6 post-transplant 2: number analyzed (Participants) | 4 | 0
  Day 6 post-transplant 2 | 31.8 (13.0) |
  Day 7 post-transplant 2: number analyzed (Participants) | 4 | 0
  Day 7 post-transplant 2 | 35.3 (12.1) |
  Month 1 (transplant 2): number analyzed (Participants) | 4 | 0
  Month 1 (transplant 2) | 28.0 (12.5) |
  Month 3 (transplant 2): number analyzed (Participants) | 4 | 0
  Month 3 (transplant 2) | 21.0 (3.6) |

19. Other Pre Specified Outcome: Serum Level of Aspartate Amino Transferase (AST)
Description: AST is commonly measured clinically as part of liver function tests.
Time Frame: Pre-transplant and at days 1-7 and months 1 and 3 post-transplant
Population: Safety population: all patients who were randomized into the study.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Reparixin | No Experimental Intervention
Number analyzed (Participants) | 6 | 3
U/L
  Pre-transplant 1 | 22.3 (14.6) | 20.0 (7.5)
  Day 1 post-transplant 1 | 30.5 (12.1) | 18.7 (7.4)
  Day 2 post-transplant 1 | 22.3 (9.2) | 27.3 (12.5)
  Day 3 post-transplant 1 | 24.7 (12.8) | 31.7 (13.4)
  Day 4 post-transplant 1 | 31.8 (9.3) | 49.0 (35.5)
  Day 5 post-transplant 1 | 60.2 (28.7) | 74.3 (26.6)
  Day 6 post-transplant 1 | 64.2 (22.1) | 64.3 (29.4)
  Day 7 post-transplant 1: number analyzed (Participants) | 5 | 3
  Day 7 post-transplant 1 | 82.0 (43.4) | 55.0 (29.7)
  Month 1 (transplant 1) | 15.5 (3.6) | 17.7 (10.0)
  Month 3 (transplant 1): number analyzed (Participants) | 4 | 0
  Month 3 (transplant 1) | 15.8 (5.0) |
  Pre-transplant 2: number analyzed (Participants) | 4 | 0
  Pre-transplant 2 | 17.0 (6.2) |
  Day 1 post-transplant 2: number analyzed (Participants) | 4 | 0
  Day 1 post-transplant 2 | 33.0 (18.7) |
  Day 2 post-transplant 2: number analyzed (Participants) | 4 | 0
  Day 2 post-transplant 2 | 21.0 (7.0) |
  Day 3 post-transplant 2: number analyzed (Participants) | 4 | 0
  Day 3 post-transplant 2 | 21.5 (5.8) |
  Day 4 post-transplant 2: number analyzed (Participants) | 4 | 0
  Day 4 post-transplant 2 | 26.8 (9.7) |
  Day 5 post-transplant 2: number analyzed (Participants) | 4 | 0
  Day 5 post-transplant 2 | 28.5 (7.5) |
  Day 6 post-transplant 2: number analyzed (Participants) | 4 | 0
  Day 6 post-transplant 2 | 23.0 (8.8) |
  Day 7 post-transplant 2: number analyzed (Participants) | 4 | 0
  Day 7 post-transplant 2 | 25.3 (10.4) |
  Month 1 (transplant 2): number analyzed (Participants) | 4 | 0
  Month 1 (transplant 2) | 17.3 (3.3) |
  Month 3 (transplant 2): number analyzed (Participants) | 3 | 0
  Month 3 (transplant 2) | 13.7 (5.0) |

20. Other Pre Specified Outcome: Change From Pre-transplant in Cytokine Levels - CXCL8
Description: Time course of inflammatory chemokines/cytokines as assessed by serum levels of CXCL8 (CXC ligand 8 [formerly interleukin (IL)-8]) (time frame: 0, 6, 12, 24, 72, 120, and 168 hours after islet infusion).
Time Frame: 6, 12, 24, 72, 120, and 168 hours post-transplant 1
Population: Safety population: all patients who were randomized into the study.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Reparixin | No Experimental Intervention
Number analyzed (Participants) | 6 | 3
pg/mL
  6 hours post-transplant | 11.0 (14.4) | 22.1 (19.0)
  12 hours post-transplant | 43.8 (45.5) | 32.9 (43.3)
  24 hours post-transplant: number analyzed (Participants) | 5 | 3
  24 hours post-transplant | 10.6 (21.8) | 11.3 (2.1)
  72 hours post-transplant | 17.3 (12.0) | 2.6 (8.5)
  120 hours post-transplant | 1.2 (8.0) | -2.2 (5.4)
  168 hours post-transplant | -6.8 (5.0) | -2.8 (1.7)

21. Other Pre Specified Outcome: Change From Pre-transplant in Cytokine Levels - CXCL1
Description: Time course of inflammatory chemokines/cytokines as assessed by serum levels of CXCL1 (time frame: 0, 6, 12, 24, 72, 120, and 168 hours after islet infusion).
Time Frame: 6, 12, 24, 72, 120, and 168 hours post-transplant 1
Population: Safety population: all patients who were randomized into the study.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Reparixin | No Experimental Intervention
Number analyzed (Participants) | 6 | 3
pg/mL
  6 hours post-transplant | -12.5 (51.8) | -31.9 (31.0)
  12 hours post-transplant | 11.8 (72.4) | -16.8 (16.2)
  24 hours post-transplant: number analyzed (Participants) | 5 | 3
  24 hours post-transplant | 1.4 (61.9) | -65.6 (127.0)
  72 hours post-transplant | 63.7 (40.7) | -51.9 (157.7)
  120 hours post-transplant | 8.7 (16.1) | -60.2 (130.6)
  168 hours post-transplant | -10.7 (65.0) | -16.3 (88.7)

22. Other Pre Specified Outcome: Change From Pre-transplant in Cytokine Levels - IL-6
Description: Time course of inflammatory chemokines/cytokines as assessed by serum levels of interleukin 6 (IL-6) (time frame: 0, 6, 12, 24, 72, 120, and 168 hours after islet infusion).
Time Frame: 6, 12, 24, 72, 120, and 168 hours post-transplant 1
Population: Safety population: all patients who were randomized into the study.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Reparixin | No Experimental Intervention
Number analyzed (Participants) | 6 | 3
pg/mL
  6 hours post-transplant | 0.5 (4.0) | 12.1 (10.6)
  12 hours post-transplant | 15.5 (20.6) | 23.4 (27.9)
  24 hours post-transplant: number analyzed (Participants) | 5 | 3
  24 hours post-transplant | 7.6 (10.7) | 2.3 (7.5)
  72 hours post-transplant | 16.3 (13.5) | 3.1 (13.3)
  120 hours post-transplant | 0.8 (5.2) | -5.6 (14.1)
  168 hours post-transplant | -2.6 (3.2) | -5.5 (8.6)

ADVERSE EVENTS:
Time Frame: Through study completion, till follow-up (up to 1 year after the second islet infusion).
Arm/Group | Reparixin | No Experimental Intervention
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 3/6 | 1/3
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reparixin (N=6) | No Experimental Intervention (N=3)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritoneal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Drug administration error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Hemorrhage (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reparixin (N=6) | No Experimental Intervention (N=3)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Infusion site pain (General disorders) | 3 (3) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0)
Hepatic haemorrhage (Hepatobiliary disorders) | 1 (1) | 0 (0)
Blood bicarbonate decreased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
Fibrin degradation product increased (Investigations) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 4 (6) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No